CLINICAL TRIAL: NCT03588000
Title: The Effect of Remote Self-monitoring of Blood Glucose (SMBG) Combined With the Promotion and Application of Internet Mobile Terminal (APP) on the Improvement of the Staged Type 2 Diabetes Mellitus (T2DM) Management and the Success Rate of Blood Glucose in the Community
Brief Title: The Effect of Remote SMBG Combined With the Application of APP on the Improvement of T2DM Management in the Community
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuwen Zhang (Other)
Responsible Party: Sponsor-Investigator, Yuwen Zhang, Principal Investigator, Ruijin Hospital
Organization: Ruijin Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16CR4020A
Record Dates: First submitted 2018-06-07; First posted 2018-07-17 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strength group (Experimental): Strengthen self-monitoring of blood glucose by Internet mobile terminal (APP)
  Interventions: Other: Strengthen self-monitoring of blood glucose
- Control group (No Intervention): Voluntary self-monitoring of blood glucose

INTERVENTIONS:
Other: Strengthen self-monitoring of blood glucose — Strengthen self-monitoring of blood glucose by Internet mobile terminal（APP）.
  Arms: Strength group

SUMMARY:
To investigate whether strengthen community diabetes patients self-monitoring of blood glucose can improve the patient's blood glucose control under Chinese guidelines for the prevention and treatment of diabetes (CDS 2017) and whether this intervention produces health and economic benefits.

DETAILED DESCRIPTION:
This project is a cohort intervention study for randomized controlled trials. Community health service centers are the main body of implementing treatment and community diabetes patients are the objects of intervention. 498 T2DM patients with poor blood glucose control (7%<HbA1c≤9.5%) from 4 different community health service centers will be randomized into two groups (strengthen group and control group). Strengthen self-monitoring of blood glucose by APP is the intervention and its duration is 12 months. Follow-up time of this study is 24 months (12 months after the intervention stopped). The diabetes treatment of patients from both groups follows Chinese guidelines (CDS 2017).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 Diabetes
* Between 18 and 79 years old
* 7.0%<HbA1c ≤ 9.5%
* Routinely uses a smart phone
* Capability of operating the designated APP
* Long-time residents in Jiading District, Shanghai, China
* Subordinated to Shanghai medical insurance
* Contracted residents of community in Jiading District, Shanghai, China
* Being cognitively able to participate
* Provision of written informed consent

Exclusion Criteria:

* Type 1 diabetes, gestational diabetes mellitus or other types of diabetes mellitus
* Currently pregnant or contemplating pregnancy within the next 24 months
* Lactating women
* Was not able to insist until the end (24 months)
* Cognitive impairment
* Migrant population

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 498 (Actual)
Dates: Start 2018-11-23 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-04-16 (Actual)

PRIMARY OUTCOMES:
absolute change in % HbA1c from baseline to 12 months | baseline to 12 months
  absolute change in glycemic control (% HbA1c) from baseline to 12 months

SECONDARY OUTCOMES:
absolute change in % HbA1c from baseline to 6 months | baseline to 6 months
  absolute change in glycemic control (% HbA1c) from baseline to 6 months
absolute change in % HbA1c from baseline at 24 months | baseline to 24 months
  absolute change in glycemic control (% HbA1c) from baseline to 24 months
change in blood glucose from baseline to 6 month | baseline to 6 months
  change in fasting and postprandial blood glucose from baseline to 6 month
change in blood glucose from baseline to 12 month | baseline to 12 months
  change in fasting and postprandial blood glucose from baseline to 12 month
change in blood glucose from baseline to 24 month | baseline to 24 months
  change in fasting and postprandial blood glucose from baseline to 24 month

OTHER OUTCOMES:
mean difference in Health-related Quality of Life Scores from baseline to 12 months | baseline to 12 months
  change in Short Form-36 (SF-36) subscale scores (Physical and Mental subscales) from baseline to 52 weeks. The SF-36 is a widely used measure of health-related quality of life.
mean difference in Health-related Quality of Life Scores from baseline to 24 months | baseline to 24 months
  change in Short Form-36 (SF-36) subscale scores (Physical and Mental subscales) from baseline to 52 weeks. The SF-36 is a widely used measure of health-related quality of life.
change in urinary albumin-to-creatinine ratio (UACR) from baseline to 12 months | baseline to 12 months
  change in urinary albumin-to-creatinine ratio (UACR) from baseline to 12 months
change in urinary albumin-to-creatinine ratio (UACR) from baseline to 24 months | baseline to 24 months
  change in urinary albumin-to-creatinine ratio (UACR) from baseline to 24 months
number of participants on specified Diabetes medications at baseline and follow-up | baseline to 12 months
  number of participants taking each of the following medications at baseline and follow-up: insulin, metformin, sulfonylurea, glinides, α-glucosidase inhibitor, glucagon-like peptide-1 (GLP-1), Thiazolidinediones (TZD), dipeptidyl peptidase IV (DPP-IV) and sodium glucose cotransporter-2 (SGLT-2).
number of participants on specified Diabetes medications at baseline and follow-up | baseline to 24 months
  number of participants taking each of the following medications at baseline and follow-up: insulin, metformin, sulfonylurea, glinides, α-glucosidase inhibitor, glucagon-like peptide-1 (GLP-1), Thiazolidinediones (TZD), dipeptidyl peptidase IV (DPP-IV) and sodium glucose cotransporter-2 (SGLT-2).
change in health economics indexes from baseline to 12 months | baseline to 12 months
  health economics indexes assessed by the number of participants taking each of the following medications at baseline and follow-up: insulin, metformin, sulfonylurea, glinides, α-glucosidase inhibitor, glucagon-like peptide-1 (GLP-1), Thiazolidinediones (TZD), dipeptidyl peptidase IV (DPP-IV) and sodium glucose cotransporter-2 (SGLT-2).
change in health economics indexes from baseline to 24 months | baseline to 24 months
  health economics indexes assessed by the number of participants taking each of the following medications at baseline and follow-up: insulin, metformin, sulfonylurea, glinides, α-glucosidase inhibitor, glucagon-like peptide-1 (GLP-1), Thiazolidinediones (TZD), dipeptidyl peptidase IV (DPP-IV) and sodium glucose cotransporter-2 (SGLT-2).

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital North, Shanghai, China